CLINICAL TRIAL: NCT02519101
Title: Impact of Continuous Noninvasive Arterial Blood Pressure Monitoring on Blood Pressure Stability During General Anaesthesia in Orthopedic Patients
Brief Title: Effects of Continuous Noninvasive Arterial Pressure Measurement on Anaesthesia
Acronym: ANIKOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Stephan Czerner, Senior Physician, Department of Anaesthesiology, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 290-15
Record Dates: First submitted 2015-08-01; First posted 2015-08-10 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Blood Pressure Stability in General Anaesthesia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continunous blood pressure monitoring (Experimental): Patients receive continuous noninvasive blood pressure monitoring in addition to intermittent monitoring
  Interventions: Device: continuous noninvasive blood pressure monitoring ClearSight-Device
- Intermittent blood pressure monitoring (No Intervention): Control group with intermittent blood pressure monitoring

INTERVENTIONS:
Device: continuous noninvasive blood pressure monitoring ClearSight-Device — Noninvasive continuous blood pressure monitoring using the volume clamp method (ClearSight-Device)
  Other Names: ClearSight-Device (Edwards)
  Arms: Continunous blood pressure monitoring

SUMMARY:
Continuous noninvasive blood pressure monitoring may help to avoid intraoperative Hypotension or Hypertension

ELIGIBILITY:
Inclusion Criteria:

* orthopedic surgery in general anaesthesia
* American Society of Anesthesiologists - Physical Status (ASA) 2 or ASA 3
* arterial Hypertension

Exclusion Criteria:

-invasive blood pressure monitoring required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Hypotensive Events in comparison between both groups | During induction and maintainance of general anaesthesia (average estimated time = 3 hours)
Dosage of Norepinephrine given to the patient to maintain blood pressure normotensive | During induction and maintainance of general anaesthesia (average estimated time = 3 hours)

SECONDARY OUTCOMES:
Incidence of acute kidney failure postoperatively | during hospital stay after surgical procedure (in average 3 days)

OTHER OUTCOMES:
mean arterial blood pressure | consecutive full hours of general anaesthesia (estimated average 3 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Anaesthesiologie am Klinikum der Universität München, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Meidert AS, Nold JS, Hornung R, Paulus AC, Zwissler B, Czerner S. The impact of continuous non-invasive arterial blood pressure monitoring on blood pressure stability during general anaesthesia in orthopaedic patients: A randomised trial. Eur J Anaesthesiol. 2017 Nov;34(11):716-722. doi: 10.1097/EJA.0000000000000690. PMID 28922340